CLINICAL TRIAL: NCT02589418
Title: Mechanisms of Acupuncture Analgesia on Experimental Dental Pain - A Randomized, Single Blinded, Sham-controlled Psychophysical Study (Phase1)
Brief Title: Mechanisms of Acupuncture Analgesia on Experimental Dental Pain - A Psychophysical Study (Phase1)
Acronym: MAC-DENT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Witt, Prof. Dr. med. Claudia M. Witt, MBA, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MAC-DENT-Psy
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Experimental Dental Pain
Keywords: Manual acupuncture; Experimental dental pain; Psychophysics; Autonomic nervous system; Subjective pain ratings
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy subjects (Experimental): All subjects participate at 3 experimental conditions (Acupuncture, Sham-Acupuncture and No Acupuncture) at 3 different days in a randomized order.
  Interventions: Procedure: Acupuncture; Procedure: Sham-Acupuncture; Procedure: No Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Needle insertion and manipulation at 4 acupuncture points (bilateral LI4, right ST6 and ST7).
  Other Names: Verum Acupuncture
Procedure: Sham-Acupuncture — Needle insertion and manipulation at 4 non-acupoints
Procedure: No Acupuncture — Control intervention: No needle insertion and manipulation

SUMMARY:
The investigators will assess the effects of manual acupuncture on experimental dental pain in 36 healthy subjects by means of subjective pain intensity ratings and pain-specific autonomic nervous system (ANS) reactions.

DETAILED DESCRIPTION:
This psychophysical and -physiological study is the first part of a two-phase project which pursues to explore how acupuncture-induced pain modulation interacts with pain-specific brain processing patterns by means of functional magnetic resonance imaging (fMRI) and by using an experimental dental pain model.

In this preceding study, the characterization of manual acupuncture effects on the experimental dental pain model will be tested under laboratory conditions and without restrictions of an fMRI-measurement in order to provide a sound foundation for the following fMRI-experiment. Pain modulating effects of the manual acupuncture intervention (4 points: needle manipulation of bilateral large-intestine 4 (LI4), stomach 6 and 7 (ST6, ST7) ipsilateral to the stimulated tooth) will be compared to sham-acupuncture (insertion and manipulation of 4 non-acupuncture points) and a control intervention (no acupuncture) which will each be performed at 3 different days in a randomized order. Intervention effects on experimental dental pain will be assessed by testing of 36 healthy volunteers by means of subjective pain intensity ratings and pain-specific ANS reactions such as electrodermal activity and heart rate/respiratory changes. Besides laying the groundwork for the following fMRI experiment, this study could provide valuable basic insights into the dynamics of the tested manual acupuncture effects and further provide important knowledge for the planning of future clinical studies encompassing dental conditions and development of acupuncture treatments.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* Written informed consent
* Fluent in German language
* Sufficient dental sensitivity for the tooth stimulation
* No acupuncture treatment in the previous 12 months
* No medical knowledge about acupuncure

Exclusion Criteria:

* Alcohol, drug, and analgesics consumption within the last 24 hours
* Complaints of diseases of the oral cavity
* Pre-existing neurological and(or psychiatric conditions
* History of severe dental pain
* Regular intake of pain medication
* History of brain injuries
* Alcohol and drug abuse
* Chronic diseases that require a permanent intake of drugs

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the - mean post-pre acupuncture intervention pain intensity rating differences - and mean post-pre control intervention (no acupuncture) rating differences | 15 minutes
Comparison of the - mean post-pre acupuncture intervention pain intensity rating differences - and mean post-pre sham-acupuncture rating differences | 15 minutes
  In case of a significant effect in outcome 1, outcome 2 will be tested using a hierarchical procedure in order to avoid multiple testing.

SECONDARY OUTCOMES:
Longer lasting effects of acupuncture on subjective intensity ratings | 50 minutes
  Besides the pre-post intervention comparisons (primary outcome), 2 additional timepoints (Total: pre-intervention, post-intervention, 15 min post-intervention, 30 min post-intervention) will be examined to test differences in temporal dynamics between the 3 intervention effects on subjective pain intensity.
Longer lasting effects of acupuncture on pain-specific changes in heart rate. | 50 minutes
  Besides the pre-post intervention comparisons (primary outcome), 2 additional timepoints (Total: pre-intervention, post-intervention, 15 min post-intervention, 30 min post-intervention) will be examined to test differences in temporal dynamics between the 3 intervention effects on pain-specific heart rate alterations.
Longer lasting effects of acupuncture on pain-specific changes in skin conductance. | 50 minutes
  Besides the pre-post intervention comparisons (primary outcome), 2 additional timepoints (Total: pre-intervention, post-intervention, 15 min post-intervention, 30 min post-intervention) will be examined to test differences in temporal dynamics between the 3 intervention effects on pain-specific skin conductance alterations.
Longer lasting effects of acupuncture on pain-specific changes in respiratory frequency. | 50 minutes
  Besides the pre-post intervention comparisons (primary outcome), 2 additional timepoints (Total: pre-intervention, post-intervention, 15 min post-intervention, 30 min post-intervention) will be examined to test differences in temporal dynamics between the 3 intervention effects on pain-specific changes in respiratory frequency.
Changes in skin conductance during the three intervention types (acupuncture, sham-Acupuncture, no acupuncture). | 10 minutes
  Comparison of changes in the skin conductance measured during the acupuncture/sham-acupuncture and no acupuncture
Changes in heart rate variability (HRV) during the three intervention types (acupuncture, sham-Acupuncture, no acupuncture). | 10 minutes
  Comparison of changes in the HRV measured during the acupuncture/sham-acupuncture and no acupuncture
Changes in respiratory frequency during the three intervention types (acupuncture, sham-Acupuncture, no acupuncture). | 10 minutes
  Comparison of changes in respiratory frequency measured during the acupuncture/sham-acupuncture and no acupuncture.
Frequency of SAEs | 1 month
  Serious adverse event (SAEs) occurrences will be recorded and their frequency will be calculated.

OTHER OUTCOMES:
Expectation towards acupuncture | 60 minutes
  Acupuncture expectation will be assessed using an acupuncture expectation questionnaire developed by the Institut for Complementary and Integrative Medicine, University Hospital Zurich
Anxiety states and traits | 60 minutes
  For the assessment of anxiety levels, the State-Trait Anxiety Inventory(STAI)(Bieling et al., 1998) questionnaire will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Clinic of Masticatory Disorders, Removable Prosthodontics, Geriatric and Special Care Dentistry Center of Dental Medicine University of Zurich, Zurich, Canton of Zurich
  - Institute for Complementary and Integrative Medicine, University Hospital Zurich, Zurich, Canton of Zurich

REFERENCES:
- [Background] Bieling PJ, Antony MM, Swinson RP. The State-Trait Anxiety Inventory, Trait version: structure and content re-examined. Behav Res Ther. 1998 Jul-Aug;36(7-8):777-88. doi: 10.1016/s0005-7967(98)00023-0. PMID 9682533
- [Derived] de Matos NMP, Pach D, Xing JJ, Barth J, Beyer LE, Shi X, Kern A, Lukic N, Ettlin DA, Brugger M, Witt CM. Evaluating the Effects of Acupuncture Using a Dental Pain Model in Healthy Subjects - A Randomized, Cross-Over Trial. J Pain. 2020 Mar-Apr;21(3-4):440-454. doi: 10.1016/j.jpain.2019.08.013. Epub 2019 Sep 12. PMID 31521794